CLINICAL TRIAL: NCT01878656
Title: Comparison of Emergence Agitation Between Sevoflurane and Desflurane Anesthesia After Orthognathic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Chongwha Baek, Chongwha Baek, M.D., Ph.D., Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Chung-Ang University Hospital
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Sevoflurane (Active Comparator): administration of sevoflurane with oxygen and nitrous oxide as same ratio of 3 L/min for maintenance of general anesthesia
  Interventions: Drug: Sevoflurane
- Desflurane (Active Comparator): administration of desflurane with oxygen and nitrous oxide as same ratio of 3 L/min for maintenance of general anesthesia
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — The investigators decrease to 1 minimal alveolar concentration(MAC) of anesthetic combination of sevoflurane and nitrous oxide, and maintain end-tidal concentration of anesthetic combination at 1 MAC until the end of surgery. At the end of surgery, sevoflurane and nitrous oxide are discontinued.
  Arms: Sevoflurane
Drug: Desflurane — The investigators decrease to 1 MAC of anesthetic combination of desflurane and nitrous oxide, and maintain end-tidal concentration of anesthetic combination at 1 MAC until the end of surgery. At the end of surgery, desflurane and nitrous oxide are discontinued.
  Arms: Desflurane

SUMMARY:
Emergence agitation is a major concern in patients undergoing orthognathic surgery. The patients may experience the sense of suffocation during emergence due to nasotracheal intubation and orofacial edema. Postoperative pain is also associated with emergence agitation. Although there is a lot of studies about emergence agitation in children, there is a few in adults, furthermore, no data about comparison of emergence agitation between sevoflurane and desflurane anesthesia in adults. Therefore, the investigators would like to compare the incidence and severity of emergence agitation between sevoflurane and desflurane anesthesia in adults after orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists(ASA) physical status classification 1 or 2 patients
* patients scheduled for orthognathic surgery

Exclusion Criteria:

* severe cardiopulmonary disease
* psychological disease
* patients who cannot understand Korean

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sevoflurane | Desflurane
Started | 72 | 72
Completed | 72 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Desflurane | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [21 to 27] | 23 [21 to 27] | 23 [21 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 50 | 96
  Male | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Emergence Agitation Using Four-point Categorical Scale
Description: The outcomes assessor will evaluate the severity of emergence agitation of participants using a four-point categorical scale. (1: calm, 2: not calm, but could be easily calmed, 3: moderately agitated or restless, 4: combative, excited, disoriented) We considered presence of emergence agitation as 3 and 4 of four-point scale.
Time Frame: Participants will be followed from the time of gas discontinuation in operating room to the time of discharge from postanesthesia care unit(PACU), an expected average of 1 hour.
Measure: Number; unit: participants
Arm/Group | Sevoflurane | Desflurane
Number analyzed (Participants) | 72 | 72
participants | 51 | 17

2. Secondary Outcome: The Time to Extubation
Description: We will evaluate the time from gas discontinuation to extubation. We will conduct an extubation when participants can show responses such as eye opening or nodding one's head to our verbal commands.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Postoperative Pain
Description: The outcomes assessor will evaluate the degree of postoperative pain using a numeric rating scale (NRS). (0 = no pain, 10 = unimaginable severe pain)
Time Frame: Participants will be followed for the duration of postanesthesia care unit (PACU) stay, an expected average of 1 hour.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Sense of Suffocation
Description: The outcomes assessor will evaluate the sense of suffocation using a numeric rating scale(NRS). (0 = no sense of suffocation, 10 = unimaginably severe sense of suffocation)
Time Frame: Participants will be followed for the duration of postanesthesia care unit (PACU) stay, an expected average of 1 hour.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sevoflurane | Desflurane
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No